CLINICAL TRIAL: NCT07097493
Title: Liposomal Bupivacaine vs Perineural Adjuvants in Adductor Canal and iPACK Blocks in Patients Undergoing Primary Total Knee Arthroplasty
Brief Title: Liposomal Bupivacaine vs Perineural Adjuvants in Adductor Canalf and iPACK Blocks in Total Knee Arthroplasty
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB00133197
Record Dates: First submitted 2025-07-24; First posted 2025-07-31 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2025-08

CONDITIONS: Knee Arthroplasty, Total
Keywords: pain; knee surgery; pain management
MeSH Terms: conditions — Pain; Agnosia | interventions — Bupivacaine; Clonidine; Epinephrine; Buprenorphine; Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Liposomal Bupivacaine (Active Comparator): randomized to liposomal bupivacaine in the adductor canal and infiltration between the popliteal artery and condyles of the knee (iPACK) block
  Interventions: Drug: Liposomal Bupivacaine
- Bupivacaine, Clonidine, Epinephrine, Buprenorphine and Dexamethasone (BPV-CEBD) (Active Comparator): randomized to bupivacaine mixed with clonidine, epinephrine, buprenorphine and dexamethasone in the adductor canal and infiltration between the popliteal artery and condyles of the knee (iPACK) block
  Interventions: Drug: Bupivacaine, Clonidine, Epinephrine, Buprenorphine and Dexamethasone (BPV-CEBD) Combination

INTERVENTIONS:
Drug: Liposomal Bupivacaine — 10 ml of 0.25% bupivacaine expanded with 133 mg (10 ml volume) of liposomal bupivacaine into both the adductor canal and iPACK blocks (total of 40 ml)
  Arms: Liposomal Bupivacaine
Drug: Bupivacaine, Clonidine, Epinephrine, Buprenorphine and Dexamethasone (BPV-CEBD) Combination — 20 ml of solution consisting of 0.25% bupivacaine, 1.667mcg/ml of clonidine, 1:400,000 epinephrine, 0.15 mg total of buprenorphine, and 2 mg total of preservative free dexamethasone which will be used in both the adductor canal block and iPACK block (total of 40 ml)
  Arms: Bupivacaine, Clonidine, Epinephrine, Buprenorphine and Dexamethasone (BPV-CEBD)

SUMMARY:
The purpose of this research study is to compare two different combinations of anesthetic medications to see which works the best in providing the longest lasting pain relief for total knee arthroplasty surgery. The drugs being used are liposomal bupivacaine compared to a combination of bupivacaine, clonidine, epinephrine, buprenorphine, and dexamethasone. Pain scores will be collected at different intervals during study participation.

DETAILED DESCRIPTION:
This double-blinded prospective randomized control trial will evaluate analgesia following total knee arthroplasty for patients who receive an adductor canal block and infiltration between the popliteal artery and condyles of the knee (iPACK) block utilizing bupivacaine with the adjuvants clonidine, epinephrine, buprenorphine and dexamethasone (BPV-CEBD), as compared to patients who receive liposomal bupivacaine (LB) for both blocks.

All patients will receive a spinal anesthetic with ropivacaine (17.5 mg) and fentanyl (10 mcg), and an adductor canal and iPACK block for analgesia. Patients randomized to the LB group will receive 10 ml of 0.25% bupivacaine expanded with 133 mg (10 ml volume) of LB into both the adductor canal and iPACK blocks (total of 40 ml). The BPV-CEBD group will receive a 20 ml of solution consisting of 0.25% bupivacaine, 1.667mcg/ml of clonidine, 1:400,000 epinephrine, 0.15 mg total of buprenorphine, and 2 mg total of preservative free dexamethasone - which will be used in both the adductor canal block and iPACK block (total of 40 ml).

On post-operative day (POD) 0, rest and movement pain scores will be collected at 4 hours and 8 hours with time "zero" being the time of the final block placement. On POD 1 and 2, questionnaires will be collected for pain scores at 0700, 1200 and 1700. Participants will be called once daily on days 3 through 7 to collect remaining secondary data, including sleep score, quality of recovery, worst daily pain score, and patient satisfaction (POD 7 only).

ELIGIBILITY:
Inclusion Criteria:

* 18-80 years of age
* Receiving primary total knee arthroplasty
* Patients receiving a spinal anesthetic with ropivacaine and fentanyl
* American Society of Anesthesiology (ASA) category 1 to 3

Exclusion Criteria:

* Revision of Total Knee Arthroplasty
* Opioid use in the prior 6 months > 40 mg oxycodone equivalents per day or long-acting opioids as determined by the Prescription Drug Monitoring Program (PDMP)
* Patients planned to receive general anesthesia
* Patients planned to receive a spinal other than ropivacaine
* History of peripheral neuropathy
* Poorly controlled diabetes (Hgb A1C >8)
* Allergies or contraindications to study medications: acetaminophen, celecoxib (including sulfa), methocarbamol, midazolam, fentanyl, bupivacaine, dexamethasone, acetaminophen, buprenorphine, NSAIDs, clonidine, epinephrine, and liposomal bupivacaine.
* Unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Pain Score with Movement | Baseline
  numerical rating scale pain score with movement utilizing the numerical rating pain score scale of 0 to 10, where 0 is no pain and 10 is the worst imaginable pain
Pain Score with Movement | Hour 4 post final block placement
  numerical rating scale pain score with movement utilizing the numerical rating pain score scale of 0 to 10, where 0 is no pain and 10 is the worst imaginable pain
Pain Score with Movement | Hour 8 post final block placement
  numerical rating scale pain score with movement utilizing the numerical rating pain score scale of 0 to 10, where 0 is no pain and 10 is the worst imaginable pain

SECONDARY OUTCOMES:
Pain Score with Rest | Hour 48 post final block placement
  numerical rating scale pain score with movement utilizing the numerical rating pain score scale of 0 to 10, where 0 is no pain and 10 is the worst imaginable pain
Pain Score with Rest | Hour 72 post final block placement
  numerical rating scale pain score with movement utilizing the numerical rating pain score scale of 0 to 10, where 0 is no pain and 10 is the worst imaginable pain
Pain Score with Movement | Hour 72 post final block placement
  numerical rating scale pain score with movement utilizing the numerical rating pain score scale of 0 to 10, where 0 is no pain and 10 is the worst imaginable pain
Highest Daily Pain Score | Postop Days 3, 4, 5, 6, 7
  numerical rating scale pain score with movement utilizing the numerical rating pain score scale of 0 to 10, where 0 is no pain and 10 is the worst imaginable pain
Cumulative Opioid Consumption | Hour 48 post final block placement
  all opioids consumed and recorded in morphine milligram equivalents (MME) for postoperative Day 2
Cumulative Opioid Consumption | Hour 72 post final block placement
  all opioids consumed and recorded in morphine milligram equivalents (MME) for postoperative Day 3
Quality of Recovery-15 Patient Survey | Postop Days 3, 4, 5, 6, 7
  quality of life questions rated on a 0-10 scale for 0=none of the time up to 10=all of the time on a daily basis; pain/nausea/vomiting/depression questions answered in a 10=none of the time down to a 0=all of the time (scales reversed on that scale)
Distance Walked | 24 hours
  distance (feet) walked during first physical therapy appointment
PROMIS Sleep Disturbance Survey | Postop Days 3, 4, 5, 6, 7
  quality of sleep rated on a scale of 0=very poor/not at all up to 5=very good/very much
Patient Satisfaction | Postop Day 7
  measured with a 5-point Likert scale 0=not satisfied at all up to 5=best level of satisfaction
Incidence of Postoperative Nausea | Up to Postop Day 7
  overall number of nausea occurrences
Incidence of Postoperative Vomiting | Up to Postop Day 7
  overall number of vomiting occurrences

CONTACTS AND LOCATIONS:
Overall Officials: Afua Gyamfi, MD, Principal Investigator — Atrium Health Wake Forest Baptist
Locations (1):
- Atrium Health Wake Forest Baptist, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No